CLINICAL TRIAL: NCT05694026
Title: Management of Dry Eye With Intense Pulsed Light in Combination With Diquafosol
Brief Title: Management of DE With IPL in Combination With DQS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPLDQS2023
Record Dates: First submitted 2023-01-10; First posted 2023-01-23 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye
Keywords: dry eye; intense pulsed light; diquafosol; tear breakup time; ocular surface disease index
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Masked examiner for all clinical assessments will not involved in the data collection or group allocation procedure for this research. The investigator will not be aware of the three groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPL+ (Experimental): Participants in the IPL+ group used DQS 1 drop 6 times/per day for four weeks along with 2 sessions of IPL, 2 weeks apart.
  Interventions: Device: Intense pulsed light; Drug: Diquafosol tetrasodium
- IPL (Experimental): IPL treatment sessions were administered once at 2- weeks interval to all participants for 4 weeks.
  Interventions: Device: Intense pulsed light
- DQS (Experimental): DQS group will be administered one drop of 3% DQS (Diquas, Santen Pharmaceutical Co., Ltd., Osaka, Japan) six times per day for 4 weeks.
  Interventions: Drug: Diquafosol tetrasodium

INTERVENTIONS:
Device: Intense pulsed light — IPL treatment intensity was chosen based on the Fitzpatrick scale as follows: Fitzpatrick scale I, II, III, 10-15 J/cm2 with a 570-nm filter.
  Other Names: IPL
  Arms: IPL; IPL+
Drug: Diquafosol tetrasodium — 3% Diquafosol tetrasodium eye drops will be used to assess its usefulness in dry eye signs and symptoms
  Other Names: Diquas
  Arms: DQS; IPL+

SUMMARY:
Intense pulsed light (IPL) has been reported to improve signs and symptoms of dry eye (DE). Additionally, meibomian gland secretion of lipids has been observed to improve through the use of IPL. Diquafosol ophthalmic solution (DQS) stimulates P2Y2 receptors on the ocular surface, which enhances mucin secretion from goblet cells. Therefore, tear film stability and hydration of the ocular surface can be achieved independent from lacrimal glands function. The purpose of this prospective study was to evaluate and compare the effects of IPL (IPL group), DQS (DQS group) and IPL in combination with DQS (IPL+ group) in participants with persistent DE. Tear film lipid layer (TFLL), non-invasive breakup time (NITBUT), tear meniscus height (TMH), corneoconjunctival staining score (CS), meibum gland (MG) function, conjunctival hyperemia (RS score), ocular surface disease index (OSDI) will be assessed and compared at baseline, day-14, and day-28.

DETAILED DESCRIPTION:
Evaporative dry eye (EDE) has been reported to be the most prevalent form of dry eye disease (DED), which is primarily caused by meibomian gland hypofunction or meibomian gland dysfunction (MGD). MGD is defined as ''a chronic, diffuse anomaly of the meibomian glands, often characterized by terminal duct blockage and/or qualitative/quantitative alterations in glandular secretion'' by the International Workshop on MGD.These glands are modified sebaceous glands that release meibum directly onto the ocular surface. Signs and symptoms of EDE and MGD can be addressed by improving the quality and quantity of meibum secretion.

Intense pulsed light (IPL) is widely used to treat dermatological conditions, and its noncoherent polychromatic light source with wide wavelength range of 500-1200 nm has been reported to stimulate facial sebaceous glands. The photothermal effect of IPL is postulated to relieve inflammation by removing aberrant surface microvasculature and enhances meibomian gland function. Furthermore, an increase in fibroblast proliferation, collagen formation and local blood flow has been associated with the application of IPL on the skin. Several studies have documented the benefits of IPL in alleviating signs and symptoms of DED on the periocular skin.

Diquafosol ophthalmic solution (DQS) is a dinucleotide polyphosphate which a purinoceptor agonist, when administered to the ocular surface, it binds to P2Y2 receptors and stimulates mucin and tear secretion. The corneal epithelium, conjunctival epithelium, lacrimal gland ductal epithelium, meibomian gland sebaceous cells, and meibomian gland ductal cells all express the P2Y2 receptor. Subsequently, enhanced secretion of mucin and tear secretion due to DQS ophthalmic solution leads to stabilization of the tear film, minimizes tear evaporation, and reduces mechanical friction thereby protecting the corneal epithelium.

The purpose of this study is to assess the management of DE by combining IPL and DQS eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Consenting participants
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease: (i) Ocular Surface Disease Index (OSDI) questionnaire ≥13, (ii) Non-invasive tear break-up (NITBUT) ≤ 5 seconds, (iii) conjunctival staining score (CS) ≥3 points. The presence of two or more criteria was used to establish a positive DE diagnosis based on the 2016 Asia Dry Eye Society criteria

Exclusion Criteria:

* A recent history (past 30 days) of topical ophthalmic medication use, including antibiotics, steroids, non-steroidal anti-inflammatory drugs, or required the chronic use of topical ophthalmic medications.
* Eyelids or intraocular tumors.
* Active allergy or infection, or inflammatory disease may prevent the subjects from completing the study at the ocular surface.
* Any structural changes in the lacrimal passage
* Glaucoma
* Diabetes or other systemic, dermatologic, or neurologic diseases that affect the health of the ocular surface.
* Use of any systemic anti-inflammatory drugs or medication that may interfere with tear production, such as antianxiety, anti-depressive, and antihistamine medications, within three months.
* Pregnancy or breastfeeding
* Contact lenses wearers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear break-up time (NIBUT) | Day-0 (baseline), day-14 and day-28
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Ocular Surface Disease Index (OSDI) | Day-0 (baseline), day-14 and day-28
  OSDI, which is a questionnaire consisting of 12 questions for evaluating the effects of dry eye syndrome on vision, ocular symptoms and any condition associated with DED. The patient will answer each question on a scale ranging from 0 to 4, with 0 indicating 'none of the time' and 4 indicating 'all of the time'. If a certain question is deemed irrelevant, it will be marked as 'not applicable (N/A)' and excluded from the analysis. The OSDI total score is calculated according to the following formula. The scale ranges from 0 to 100, with higher scores representing more severe cases of dry eye syndrome.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined

SECONDARY OUTCOMES:
Fluorescein and lissamine conjunctival and cornea staining (CFS) | Day-0 (baseline), day-14 and day-28
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Meibomian gland function and secretion quality | Day-0 (baseline), day-14 and day-28
  Meibum quality will be assessed under a slit-lamp: Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum)
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Tear Film Lipid Layer Score (TFLL) | Day-0 (baseline), day-14 and day-28
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan). The results will be graded as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Tear meniscus height (TMH) | Day-0 (baseline), day-14 and day-28
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded.
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.
Conjunctival hyperemia (RS score) | Day-0 (baseline), day-14 and day-28
  Conjunctival hyperemia (RS score) will be assessed by Keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 (normal) to 4.0 (severe).
  * Changes at day-14 and day-28 will be compare with baseline measurements.
  * Comparison between groups at baseline, day-14 and day-28 will also be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, MD, PhD, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: The Steering Committee will write and submit the report for publication at the end of the study
Access Criteria: Use in clinical studies

REFERENCES:
- [Result] Ma J, Pazo EE, Zou Z, Jin F. Prevalence of symptomatic dry eye in breast cancer patients undergoing systemic adjuvant treatment: A cross-sectional study. Breast. 2020 Oct;53:164-171. doi: 10.1016/j.breast.2020.07.009. Epub 2020 Aug 5. PMID 32836200
- [Result] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Result] Bron AJ, Tiffany JM. The contribution of meibomian disease to dry eye. Ocul Surf. 2004 Apr;2(2):149-65. doi: 10.1016/s1542-0124(12)70150-7. PMID 17216085
- [Result] Chhadva P, Goldhardt R, Galor A. Meibomian Gland Disease: The Role of Gland Dysfunction in Dry Eye Disease. Ophthalmology. 2017 Nov;124(11S):S20-S26. doi: 10.1016/j.ophtha.2017.05.031. PMID 29055358
- [Result] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Result] Raulin C, Greve B, Grema H. IPL technology: a review. Lasers Surg Med. 2003;32(2):78-87. doi: 10.1002/lsm.10145. PMID 12561039
- [Result] Heymann WR. Intense pulsed light. J Am Acad Dermatol. 2007 Mar;56(3):466-7. doi: 10.1016/j.jaad.2006.10.031. No abstract available. PMID 17317488
- [Result] Liu R, Rong B, Tu P, Tang Y, Song W, Toyos R, Toyos M, Yan X. Analysis of Cytokine Levels in Tears and Clinical Correlations After Intense Pulsed Light Treating Meibomian Gland Dysfunction. Am J Ophthalmol. 2017 Nov;183:81-90. doi: 10.1016/j.ajo.2017.08.021. Epub 2017 Sep 6. PMID 28887117
- [Result] Baumler W, Vural E, Landthaler M, Muzzi F, Shafirstein G. The effects of intense pulsed light (IPL) on blood vessels investigated by mathematical modeling. Lasers Surg Med. 2007 Feb;39(2):132-9. doi: 10.1002/lsm.20408. PMID 17066482
- [Result] Jeng SF, Chen JA, Chang LR, Chen CC, Shih HS, Chou TM, Chen HF, Feng GM, Yang CH. Beneficial Effect of Intense Pulsed Light on the Wound Healing in Diabetic Rats. Lasers Surg Med. 2020 Jul;52(6):530-536. doi: 10.1002/lsm.23183. Epub 2019 Nov 24. PMID 31763712
- [Result] Cao Y, Huo R, Feng Y, Li Q, Wang F. Effects of intense pulsed light on the biological properties and ultrastructure of skin dermal fibroblasts: potential roles in photoaging. Photomed Laser Surg. 2011 May;29(5):327-32. doi: 10.1089/pho.2010.2867. Epub 2011 Mar 25. PMID 21438701
- [Result] Chen Y, Li J, Wu Y, Lin X, Deng X, Yun-E Z. Comparative Evaluation in Intense Pulsed Light Therapy Combined with or without Meibomian Gland Expression for the Treatment of Meibomian Gland Dysfunction. Curr Eye Res. 2021 Aug;46(8):1125-1131. doi: 10.1080/02713683.2020.1867750. Epub 2021 Jan 18. PMID 33342317
- [Result] Pazo EE, Huang H, Fan Q, Zhang C, Yue Y, Yang L, Xu L, Moore JE, He W. Intense Pulse Light for Treating Post-LASIK Refractory Dry Eye. Photobiomodul Photomed Laser Surg. 2021 Mar;39(3):155-163. doi: 10.1089/photob.2020.4931. Epub 2020 Dec 8. PMID 33296261
- [Result] Kulkarni AA, Trousdale MD, Stevenson D, Gukasyan HJ, Shiue MH, Kim KJ, Read RW, Lee VH. Nucleotide-induced restoration of conjunctival chloride and fluid secretion in adenovirus type 5-infected pigmented rabbit eyes. J Pharmacol Exp Ther. 2003 Jun;305(3):1206-11. doi: 10.1124/jpet.103.049221. Epub 2003 Mar 20. PMID 12649304
- [Result] Dota A, Sakamoto A, Nagano T, Murakami T, Matsugi T. Effect of Diquafosol Ophthalmic Solution on Airflow-Induced Ocular Surface Disorder in Diabetic Rats. Clin Ophthalmol. 2020 Apr 1;14:1019-1024. doi: 10.2147/OPTH.S242764. eCollection 2020. PMID 32280196
- [Result] Jumblatt JE, Jumblatt MM. Regulation of ocular mucin secretion by P2Y2 nucleotide receptors in rabbit and human conjunctiva. Exp Eye Res. 1998 Sep;67(3):341-6. doi: 10.1006/exer.1998.0520. PMID 9778415
- [Result] Tanioka H, Kuriki Y, Sakamoto A, Katsuta O, Kawazu K, Nakamura M. Expression of the P2Y(2) receptor on the rat ocular surface during a 1-year rearing period. Jpn J Ophthalmol. 2014 Nov;58(6):515-21. doi: 10.1007/s10384-014-0342-4. Epub 2014 Sep 2. PMID 25179431
- [Result] Cowlen MS, Zhang VZ, Warnock L, Moyer CF, Peterson WM, Yerxa BR. Localization of ocular P2Y2 receptor gene expression by in situ hybridization. Exp Eye Res. 2003 Jul;77(1):77-84. doi: 10.1016/s0014-4835(03)00068-x. PMID 12823990
- [Derived] Chen J, Qin G, Li L, Qi Y, Che H, Huang H, Xia Y, Zhang Q, Wu Y, Yang L, Moutari S, Moore JE, Xu L, He W, Yu S, Pazo EE, He X. Protocol for a parallel assignment prospective, randomised, comparative trial to evaluate the safety and efficacy of intense pulsed light (IPL) combined with 3% diquafosol (DQS) ophthalmic solution in dry eye syndrome. BMJ Open. 2023 Aug 29;13(8):e073055. doi: 10.1136/bmjopen-2023-073055. PMID 37643847
- [Derived] Chen J, Qin G, Li L, Qi Y, Xia Y, Zhang Q, Wu Y, You Y, Yang L, Guo N, Moutari S, Moore JE, Bu S, Xu L, He W, Yu S, Pazo EE, He X. The Combined Impact of Intense Pulsed Light Combined and 3% Diquafosol Ophthalmic Solution on Evaporative Dry Eye: A Randomized Control Study. Ophthalmol Ther. 2023 Dec;12(6):2959-2971. doi: 10.1007/s40123-023-00784-z. Epub 2023 Aug 17. PMID 37589932